CLINICAL TRIAL: NCT04819399
Title: Phase I, Open Label, Dose Escalating Study to Investigate Safety and Tolerability of Intravesical Application of Trifunctional Anti-EPCAM x Anti-CD3 Antibody Catumaxomab in Patients With Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Investigation of Safety and Tolerability of Catumaxomab in Patients With NMIBC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lindis Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CATUNIBLA; 2019-002850-22 (EudraCT Number)
Record Dates: First submitted 2021-03-18; First posted 2021-03-29 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Non Muscle Invasive Bladder Cancer; NMIBC; Catumaxomab; Intravesical
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catumaxomab (Experimental): intravesical Catumaxomab instillation
  Interventions: Drug: Catumaxomab

INTERVENTIONS:
Drug: Catumaxomab — Procedure: 6 weekly intravesical administration at each dose level; 3 sequential cohorts consisting of 3 patients (part I)
  1. cohort 50 µg
  2. cohort 70 µg
  3. cohort 100 µg
  Part II will be treated at recommended dose

SUMMARY:
The purpose of the study is to investigate the safety, tolerability, and preliminary efficacy of the monoclonal bispecific trifunctional antibody Catumaxomab in patients with non-muscle invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
The present Phase I dose escalation study (CATUNIBLA) in patients with non-muscle invasive bladder cancer (NMIBC) of high and intermediate risk for progression aims at investigating the therapeutic potential of Catumaxomab applied as intravesical instillation. Catumaxomab is an intact trifunctional bispecific monoclonal antibody and has the molecular targets EpCAM and CD3. It mediates antibody-dependent cellular cytotoxicity against human epithelial tumor cells including bladder cancer.

The study consists of two parts: Part I is dose finding and will investigate 3 sequential cohorts consisting of 3 patients to be enrolled at the specified dose levels. After determination of the dose for Part II an additional number (n=X) of patients will be included at this dose level. Part I and part II have a screening period, 6 week treatment phase and a follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

Patients will be enrolled in this Phase I study only if they meet all of the following criteria:

* Male or non-pregnant, non-breastfeeding female, age 18 years or older at date of consent.
* Any of the following histologically confirmed non-muscle invasive urothelial carcinoma of the bladder:

High-risk tumors according to EAU guidelines:

* pT1
* G3 HG tumors
* CIS
* Multiple, recurrent and large (>3cm) pTa G1-G2 LG tumors (all features must be present)

  * Patients of the subgroup of highest risk tumours (T1G3/HG associated with concurrent bladder CIS, multiple- and/or large T1G3/HG and/or recurrent T1G3/HG, T1G3/HG with CIS in the prostatic urethra, some forms of variant histology of urothelial carcinoma, lymphovascular invasion) will be only enrolled if they have already failed BCG-treatment or they cannot tolerate it and are ineligible or refuse cystectomy. In the Part II of the study a minimal expression of EpCAM in the tumor tissue may be required, based on preliminary evidence from the Part I of the study
  * Previous therapies must be discontinued at least 2 weeks prior to administration of Catumaxomab and all treatment related toxicities must have resolved or decreased to common toxicity criteria (CTCAE) grade 1.
  * Time period from primary resection to antibody treatment start must be at least one week and should not exceed 2 weeks.
  * Any investigational agent must be discontinued at least 4 weeks or 5 half-lives, whichever is longer, prior to antibody treatment start.
  * Female patients of child-bearing potential (for definition refer to section 14.3)must:
* have negative serum pregnancy test prior to study treatment to rule out pregnancy.
* Use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), true sexual abstinence or vasectomized partner from the time of signing the informed consent through 2 weeks after the last study drug treatment.

  * All sexually active patients agree to use barrier contraception (i.e., condoms) while receiving study treatment and for 2 weeks following their last dose of study treatment.
  * Adequate organ function, as defined by the following criteria:
* Aspartate aminotransferase / serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase / serum glutamic pyruvate transaminase (ALT/SGPT) ≤ 3.0 x upper limit of normal (ULN);
* Total serum bilirubin ≤ 1.5 x ULN (CTCAE Grade ≤ 1);
* Serum creatinine ≤ 1.5 x ULN; or a creatinine clearance ≥40 ml/min
* Alkaline phosphatase < 2.5 x ULN

  • Adequate hematological, liver and kidney function:
* Hemoglobin ≥8.0 g/dL;
* Absolute neutrophil count ≥1500/mm3;
* Platelets ≥75,000mm3(= 75 G/l)
* Activated Partial thromboplastin time (aPTT) within limits of normal • Signed and dated informed consent/assent form

Exclusion Criteria:

Patients will not be enrolled in this Phase I study if they meet any of the following criteria:

* The female patient is pregnant, lactating or breastfeeding or has a positive serum pregnancy test during the screening period.
* Low risk or intermediate risk tumors according to EAU guidelines
* History or signs (obstruction of upper urinary tract or cross hematuria in the ureteral orifice) of urethral or upper tract transitional cell carcinoma (TCC). Patients with T1 disease of the bladder must have no evidence of upper or lower tract disease or a more advanced stage of disease by either computed tomography (CT) urography or magnetic resonance imaging (MRI) urography of the abdomen and pelvis performed within 8 weeks before the first application of study treatment. If intravenous contrast medium for CT and MRI is contraindicated, retrograde ureteropyelography, or CT or MRI without intravenous contras tmedia may be performed.
* Patients with hydronephrosis.
* Any intravesicular or other chemotherapy treatment within 2 weeks or any investigational agent within 4 weeks or 5 half-lives of the agent whatever is longer prior to the initial dose of study drug
* History of recurrent severe urinary tract infections (UTIs) per investigator judgment.
* Active, uncontrolled impairment of the urogenital, renal, hepatobiliary, cardiovascular, gastrointestinal, neurologic or hematopoietic systems which, in the opinion of the investigator, would predispose the patient to the development of complications from the administration of intravesical therapy.
* A diagnosis of another malignancy within 2 years before the first dose of study treatment, except for superficial skin cancer or localized solid tumors deemed cured by surgery and not treated with systemic anticancer therapy and not expected to require anticancer therapy within the next 2 years i.e., while the patient may be taking study treatment or is in the follow up period of this study.

  * Patients with a history of cancer who have completed treatment and are free from disease since at least 5 years can be enrolled.
  * Patients with low-risk prostate cancer, e.g.:
  * Clinically localized disease (≤T2a) and
  * Gleason score ≤6 (3+3) and
  * Serum PSA <10 ng/ml undergoing active surveillance may be enrolled with agreement of the sponsor.
* Patients who cannot tolerate intravesical administration or intravesical surgical manipulation (cystoscopy, biopsy) due to the presence of serious comorbid condition(s) (e.g., uncontrolled cardiac or respiratory disorders).
* Known hypersensitivity to Catumaxomab and its analogues in general, or to any other component of the study drug formulation.
* Documented acute or chronic infection including known hepatitis B or C or HIV infection or other concurrent non-malignant co morbidities such as unstable or uncontrolled pectoral angina, myocardial infarction during the last 6 months, valvular heart disease that requires treatment, acute myocarditis or congestive heart failure (CHF) (New York Heart Association (NYHA) III or IV).
* Any concurrent chemotherapy, radiotherapy (except for local radiation therapy for bone metastasis), immunotherapy or corticoid therapy.

Any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the study as judged by the investigator.

* Participation in any of the following types of clinical studies either concurrently or within the previous 28 days or within 5 half-lives of any investigational pharmacologic agents, whichever is longer: pharmacologic agents or imaging materials, including dyes, investigational surgical techniques or devices. Participation in studies of psychology, or socioeconomic issues is allowed.
* Unwilling or unable to follow protocol requirements.
* Legal incompetence or limited legal competence, or detainment in an institution due to official or legal reasons
* Involvement in the conduct and/or the design of the study (applies to sponsor's staff or staff in treating centres)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose escalation phase to evaluate DLT incidence | approximately 1 year after study start
  Dose Limited Toxicity
Incidence and severity of treatment related adverse events | approximately 2.5 years after study start
  Incidence and severity of treatment related adverse events during intravesical instillation with catumaxomab are observed according to NCI CTCAE, Version 5.0

SECONDARY OUTCOMES:
Anti-drug antibodies (ng/ml) | approximately 2.5 years after study start
  the incidence of ADA (anti-drug antibodies to catumaxomab by intravesical instillation in serum
Cytokines (pg/mL) | approximately 2.5 years after study start
  cytokines (pg/mL)
Number of EpCAM-positive tumor cells in the urine | approximately 2.5 years after study start
  • number of EpCAM-positive tumor cells in the urine
Number of immune cells in the urine | approximately 2.5 years after study start
  • number of immune cells in the urine
Cmax (ng/ml) | approximately 2.5 years after study start
  PK parameter of Catumaxomab is Cmax (ng/ml)
Cmin (ng/ml) | approximately 2.5 years after study start
  PK parameters of Catumaxomab is Cmin (ng/ml)
Tmax (hours) | approximately 2.5 years after study start
  PK parameter of Catumaxomab is Tmax (hours)
AUC (day * ng/ml) | approximately 2.5 years after study start
  PK parameters of Catumaxomab AUC (day * ng/ml)
t1/2 (days) | approximately 2.5 years after study start
  PK parameter of Catumaxomab t1/2 (days)
Antitumor activity | approximately 2.5 years after study start
  antitumor activities is assessed by cystoscopy and biopsy/or resection at EoT (day 43) and all follow up visits and measures and documents tumor size, tumor localization, tumor numbers and morphological criteria
Complete response | approximately 2.5 years after study start
  Complete response will be defined as no histological evidence of disease at 3-monthly evaluations
Recurrence-free interval | approximately 2.5 years after study start
  recurrence-free interval is evaluated following the catumaxomab treatment in the follow up phase 3 month to 2 years
Local progression free interval | approximately 2.5 years after study start
  local progression free interval is evaluated following the catumaxomab treatment in the follow up phase 3 month to 2 years
Identification and quantification of tumor cells in urine | approximately 2.5 years after study start
  this is evalulated at screening and in the course of the study
EpCAM expression | approximately 2.5 years after study start
  Evaluation of potential and predictive EpCAM expression and relative Lymphocytes count can be correlated with outcome

CONTACTS AND LOCATIONS:
Overall Officials: R Oberneder, MD, Principal Investigator — Urologische Klinik München-Planegg
Locations (1):
- Urologie Planegg, München, Germany